CLINICAL TRIAL: NCT04771871
Title: Treatment Response and microRNA Profiles in Triple Negative Breast Cancer Patients Receiving Standard Chemotherapy
Brief Title: MicroRNA Profiles in Triple Negative Breast Cancer
Acronym: TARMAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital, Ibadan (Other)
Collaborators: Lagos State University (Other); Obafemi Awolowo University Teaching Hospital (Other); University of Chicago (Other); University of Lagos, Nigeria (Other); University of Ibadan (Other)
Responsible Party: Principal Investigator, Atara Ntekim, Study Principal Investigator, University College Hospital, Ibadan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UI-ROD-OCTU02
Record Dates: First submitted 2021-02-14; First posted 2021-02-25 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast cancer; neoadjuvant treatment; microRNA; circulating tumor cells
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Epirubicin; Paclitaxel; Carboplatin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: This is a one-stage phase II study with a single arm design. All patients will receive 4 cycles of epirubicin + cyclophosphamide followed by paclitaxel +carboplatin for four cycles in the neo-adjuvant setting. Those with clinical response (assessed via breast ultrasound), will undergo surgery. After surgery, all patients who achieve pCR will undergo radiotherapy. Patients with pathological incomplete response or stable disease may have additional chemotherapy at the discretion of the managing physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epirubicin-Cyclophosphamide plus Paclitaxel- Carboplatin (Experimental): Epirubicin 60mg/m2 with cyclophosphamide 600/m2 every three weeks for four courses followed by paclitaxel 120mg/m2 and carboplatin 6 AUC every three weeks for four courses
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Epirubicin — Epirubicin is an antitumor antibiotics with good activity on breast cancer. It has less cardiotoxic effect than doxorubicin
  Other Names: Pharmorubicin; Taxol; Paraplatin; Cytoxan
Drug: Cyclophosphamide — Cyclophosphamide is a cytoxic drug indicated for the treatment of many malignancies including breast cancer
  Other Names: Cytoxan
Drug: Paclitaxel — Paclitaxel is a taxane chemotherapy agent indicated for the treatment of many cancers including breast cancer. It can be used alone or in combination with other drugs
  Other Names: Taxol
Drug: Carboplatin — Carboplatin is a platinum compound indicated for the treatment of many types of malignancies including breast cancer
  Other Names: Carboplat; Paraplatin

SUMMARY:
Triple negative breast cancer (TNBC) is an aggressive disease with higher proportion of Blacks affected and in younger age groups. There is no targeted therapy unlike other types of breast cancer such as hormone positive and Human Epidermal Growth factor 2 (HER2) positive subtypes. Chemotherapy is therefore the main choice of systemic treatment with rapid development of resistance in most cases. At present, there is no blood test to monitor treatment response and disease relapse. This one-stage phase II study with a single arm design will determine the response rate of standard chemotherapy using Epirubicin (60mg/m2), Cyclophosphamide (600mg/m2) , Paclitaxel (120mg/m2) and Carboplatin (6AUC) in TNBC patients. We will measure the blood level of microRNA molecules and circulating tumor DNA during and after treatment to test if changes can be used to indicate drug failure in these patients. Disease status and tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guidelines while toxicity will be assessed using CTCAE v5). The trial will be conducted as per the International Council on Harmonisation Good Clinical Practice (ICH GCP) Guidelines E6 (R1) and other applicable guidelines

DETAILED DESCRIPTION:
Triple negative subtype of breast cancer (TNBC), accounts for about 55% of all breast cancer among indigenous blacks, such as Nigerians, and younger women are more susceptible Patients with TNBC generally experience a more aggressive clinical course with faster disease progression and poorer overall survival. There is no targeted treatment available beyond conventional cytotoxic chemotherapy . Unfortunately, standard chemotherapy is only effective in about 40% of patients with pathological complete response (pCR) achieved only in 20%-30% . Local relapse occurs early. Therefore, chemo-resistance is the main cause of chemotherapeutic failure and leads to suboptimal response rates . There are no biomarkers of response for close monitoring of TNBC patients to identify chemotherapy failure early. This one-stage phase II study with a single arm is designed to assess the response rate and toxicity of Epirubicin-Cyclophosphamide with Paclitaxel-Carboplatin (ECPC) and examine the potential of using circulating microRNa and circulating tumor cells as a surrogate marker of chemotherapy resistance in Nigerian women with triple negative breast cancer. A total of 42 patients will be enrolled into the trial. Each participant will receive Epirubicin (60mg/m2), Cyclophosphamide (600mg/m2) , Paclitaxel (120mg/m2) and Carboplatin (6AUC) . Blood microRNA and circulating tumor DNA will be determined before and after therapy. Tumor response will be measured by breast ultrasound and described using RECIST criteria while toxicity will be graded using CTCAE criteria. Quality of life (QoL) of participants while on chemotherapy will also be assessed using EORTC quality of life questionnaire - (General and Breast cancer specific).

ELIGIBILITY:
Inclusion Criteria:

1. Women ages of 18 to 70 years old
2. Women who give informed consent for the study
3. Biopsy-accessible breast tumor of significant size for core needle biopsy/ultrasound measurable (≥ 2cm)
4. Patients with histologically confirmed carcinoma of the female breast with triple negative status by immuno-histochemistry (IHC)
5. Clinical stages IIA -IIIC (AJCC 2009)
6. Chemotherapy-naïve patients (for this malignancy)
7. Performance status: Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Non-pregnant and not nursing. Women of childbearing potential must take the pregnancy test and must commit to receive Leuteinizing Hormone Realising Hormone (LHRH) agonist Zoladex (goserelin) for two years starting from the commencement of the study medications
9. Required Initial Laboratory Data. Adequate hematologic, renal and hepatic function, as defined by each of the following:

1. Granulocyte ≥ 1,500/μL 2. Platelet count ≥ 100,000/μL 3. Absolute neutrophil count (ANC) ≥ l500/μL 4. Hemoglobin ≥ 10g/dL 5. Bilirubin ≤ 1.5 x upper limit of normal 6. SGOT and SGPT < 2.5 x upper limit of normal 7. Creatinine within institutional normal limits or glomerular filtration rate ≥ 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) (CKD EPI) equation (see http://mdrd.com/ for calculator) 10. Echocardiogram (ECHO): Baseline left ventricular ejection fraction of ≥ 55%

Exclusion Criteria:

1. Pregnant or lactating women. Women of childbearing potential not using a reliable and appropriate contraceptive method. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
2. Patients with distant metastasis (brain and/or visceral metastasis)
3. Serious, uncontrolled, concurrent infection(s).
4. Treatment for other carcinomas within the last 5 years, except non-melanoma skin cancer and treated cervical carcinoma in-situ (CCIS)
5. Participation in any investigational drug study within 4 weeks preceding the start of study treatment
6. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation including but not limited to chronic or active infection, HIV-positive patient, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled Diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Bilogical females will be used. This is because female breast are larger with measurable tumor sizes. In addition, microRNA expression will be more uniform in females for this study
Enrollment: 42 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving pathological complete response (pCR) at surgery following neoadjuvant treatment with epirubicin + cyclophosphamide every three weeks for four cycles followed by paclitaxel + carboplatin every three weeks for four cycles | 4 - 6 months from commencement of chemotherapy. (Surgery will be performed within 4-6 weeks after completion of chemotherapy
  Percentage of participants achieving pathological complete response (pCR) at surgery
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From the date of commencement of chemotherapy till date of first documentation of adverse event up to 60 months or withdrawal or death from any cause or which ever occurs first.
  Percentage of participants experiencing grades 3 and 4 hematological, gastro-intestinal, neurological and cardiovascular toxicities.

SECONDARY OUTCOMES:
Number of Participants without disease for 2 , 5 and 10 years respectively | From date of first dose of study drug treatment up to a maximum of 120 months years.
  Invasive Disease Free Survival (iDFS )
Change in quality of life (QoL) score of patients from baseline using the EORTC quality of life questionnaire during chemotherapy and at study completion | From date of commencement of study medications up to 60 months
  The various domains of QoL over time and the changes from baseline using the validated European Organization for Research and Treatment of Cancer (EORTC)) QoL instrument (global and breast module).

OTHER OUTCOMES:
The serum levels of circulating microRNAs during chemotherapy in TNBC. To explore mechanisms of resistance to chemotherapy in Nigerian women with TNBC | From date of commencement of chemotherapy up to 24 weeks
  The fold change in serum levels of miRNA during chemotherapy will be determine in TNBC patients before and during each course of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo I. Olopade, Study Chair — University of Chicago; Atara Ntekim, Principal Investigator — University of Ibadan
Locations (4):
- Nigeria (4):
  - Obafemi Awolowo University Teaching Hospital, Ile-Ife, Oshun
  - University College Hospital, Ibadan, Oyo State
  - Lagos State University Teaching Hospital, Lagos
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification. The data will be deposited with the journal as supplementary data. Access will be as per journals policy
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication. No end date
Access Criteria: As per publishing Journal's policy

REFERENCES:
- [Background] Adalsteinsson VA, Ha G, Freeman SS, Choudhury AD, Stover DG, Parsons HA, Gydush G, Reed SC, Rotem D, Rhoades J, Loginov D, Livitz D, Rosebrock D, Leshchiner I, Kim J, Stewart C, Rosenberg M, Francis JM, Zhang CZ, Cohen O, Oh C, Ding H, Polak P, Lloyd M, Mahmud S, Helvie K, Merrill MS, Santiago RA, O'Connor EP, Jeong SH, Leeson R, Barry RM, Kramkowski JF, Zhang Z, Polacek L, Lohr JG, Schleicher M, Lipscomb E, Saltzman A, Oliver NM, Marini L, Waks AG, Harshman LC, Tolaney SM, Van Allen EM, Winer EP, Lin NU, Nakabayashi M, Taplin ME, Johannessen CM, Garraway LA, Golub TR, Boehm JS, Wagle N, Getz G, Love JC, Meyerson M. Scalable whole-exome sequencing of cell-free DNA reveals high concordance with metastatic tumors. Nat Commun. 2017 Nov 6;8(1):1324. doi: 10.1038/s41467-017-00965-y. PMID 29109393
- [Background] Aebi S, Davidson T, Gruber G, Cardoso F; ESMO Guidelines Working Group. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2011 Sep;22 Suppl 6:vi12-24. doi: 10.1093/annonc/mdr371. No abstract available. PMID 21908498
- [Background] Kaufmann M, von Minckwitz G, Mamounas EP, Cameron D, Carey LA, Cristofanilli M, Denkert C, Eiermann W, Gnant M, Harris JR, Karn T, Liedtke C, Mauri D, Rouzier R, Ruckhaeberle E, Semiglazov V, Symmans WF, Tutt A, Pusztai L. Recommendations from an international consensus conference on the current status and future of neoadjuvant systemic therapy in primary breast cancer. Ann Surg Oncol. 2012 May;19(5):1508-16. doi: 10.1245/s10434-011-2108-2. Epub 2011 Dec 23. PMID 22193884
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361